CLINICAL TRIAL: NCT03186846
Title: Influence of Volume Optimisation on Cognitive Function in Major Abdominal Surgery
Brief Title: Volume Optimisation and Cognitive Function in Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Alenka Spindler-Vesel, MD, PhD, Head of anaesthesiology department for abdominal surgery, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KME 21/11/16
Record Dates: First submitted 2017-05-18; First posted 2017-06-14 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Cognitive Decline
Keywords: cognitive decline; hemodynamic monitoring; LIDCO; INVOS; BIS; brain injury biomarkers
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multimodal monitoring (Active Comparator): LiDCO Rapid, unilateral INVOS and unilateral BIS monitors will be applied. Should there be pre-existing carotid stenosis, INVOS sensor will be applied on the same side. In case of pre-existing cerebral pathology, the INVOS sensor will be applied to the contralateral side. Baseline values of nominal stroke index (SI), cardiac index (CI), BIS, mean arterial pressure (MAP) and regional oxygen saturation (rSO2) will be recorded. Basal rSO2 will be recorded prior to preoxygenation which raises the value. Before the induction, up to 250ml of balanced crystalloid solution will be administered. These will include antibiotics solvents and other pre-induction i.v. therapy.
  Interventions: Device: multimodal monitoring
- placebo (Active Comparator): No multimodal monitoring will be applied in control group.
  Interventions: Device: placebo

INTERVENTIONS:
Device: multimodal monitoring — LiDCO Rapid, unilateral INVOS and unilateral BIS monitors will be applied. Should there be pre-existing carotid stenosis, INVOS sensor will be applied on the same side. In case of pre-existing cerebral pathology, the INVOS sensor will be applied to the contralateral side. Baseline values of nominal stroke index (SI), cardiac index (CI), BIS, mean arterial pressure (MAP) and regional oxygen saturation (rSO2) will be recorded. Basal rSO2 will be recorded prior to preoxygenation which raises the value. • Before the induction, up to 250ml of balanced crystalloid solution will be administered. These will include antibiotics solvents and other pre-induction i.v. therapy.
  Other Names: LiDCO Rapid, unilateral INVOS, unilateral BIS
  Arms: multimodal monitoring
Device: placebo — Before the induction, up to 250ml of balanced crystalloid solution will be administered. These will include antibiotics solvents and other pre-induction i.v. therapy.
  Arms: placebo

SUMMARY:
In the last 25 years, there has been a lot of attention directed on reducing perioperative morbidity and mortality by improving intraoperative monitoring and hemodynamic optimisation of patients. Advanced monitoring devices and new parameters have shifted the focus of anaesthesia management from macro- to micro circulation with the emphasis on the determinants of oxygen delivery and tissue oxygenation. There is increasing evidence that long-term outcome is improved by goal-directed optimisation of hemodynamic parameters (optimisation of stroke volume and cardiac output by fluids and inotropic and vasoactive drugs). Besides, new monitoring possibilities (depth of anaesthesia and cerebral and tissue oxygenation monitors) and adherence to protocols have proved beneficial in reducing morbidity cognitive dysfunction.

However, questions are raised what the optimal goals (healthy population derived normal values, preoperative values, maximal values, restrictive fluid management) should be. Secondly, all new methods were used separately and there is a lack of studies to show the effect of combined (multimodal) monitoring on occurrence of cognitive dysfunction. All gathered data indicate that the combined use of new methods with adherence to an appropriate protocol might radically improve the perioperative management and outcome of high-risk surgical patients.

The present study tests the hypothesis that intraoperative multimodal monitoring with hemodynamic optimisation, BIS-guided anaesthesia and maintenance of optimal cerebral oxygen saturation will reduce cognitive dysfunction.

DETAILED DESCRIPTION:
BACKGROUND There is increasing evidence that intraoperative aesthetic management influences outcomes. (5). Besides this the occurrence of low MAP, low minimum alveolar concentration (MAC) and low bispectral index (BIS) increased hospital stay and mortality.

Conventional intraoperative monitoring can result in occult low levels of blood flow and oxygen delivery that lead to complications that only occur days or weeks following surgery and give false re-assurance to the anaesthetist that he or she is doing a "good job". Advanced monitoring devices and new parameters have shifted the focus of anaesthesia management from macro- to microcirculation with the emphasis on the determinants of oxygen delivery and tissue oxygenation. There are more and more trials showing that introduction of new monitors and treatment protocols with predefined treatment limits or targets (goal-directed optimisation of hemodynamic parameters) improves long-term patient outcome and reduces morbidity and mortality by over 50%. Several studies have shown benefit when individualised; targeted oxygen delivery algorithms incorporating both fluid resuscitation and vasoactive drugs were used with high-risk surgical patients. The measurement of regional cerebral oxygen saturation can predict cognitive dysfunction after cardiac surgery. BIS monitoring facilitates anaesthetic titration, and reduced anaesthetic exposure and decreased the risk of postoperative cognitive dysfunction. There is reduction in strokes, less mechanical ventilation and shorter length of stay (LOS) with the use of INVOS.

However, all new methods have been studied separately and there is a lack of studies to show the effect of combined (multimodal) monitoring on mortality and occurrence of complications, including cognitive decline. All gathered data indicate that the combined use of new methods (assessment of fluid status, depth of anaesthesia and tissue oxygenation) with adherence to appropriate protocol might radically improve perioperative management and outcome of high-risk surgical patients.

Besides, questions are raised what the optimal goals (healthy population derived normal values, preoperative values, maximal values) should be. Lately, studies have shown that optimising cardiac output and oxygen delivery to higher (supra-normal) values intra- and postoperatively did not affect post-operative complications rate, intensive care unit stay or hospital length of stay. Probably the target should be maintaining patient's blood flow and oxygen delivery at preinduction levels. The question was also raised in fluid management. Liberal approach can lead to oedema of the intestines and other tissues, which may be responsible for poor tissue healing and other complications. In abdominal surgery, protocol-based fluid restriction reduced the incidence of perioperative complications such as cardiopulmonary events and disturbances of bowel motility while improving wound and anastomotic healing and reducing hospital stay in comparison to liberal fluid management. One of the trials has shown 52% lower rate of major postoperative complications in restrictive group than in the conventional group.

HYPOTHESIS The present study tests the hypothesis that intraoperative multimodal monitoring with hemodynamic optimisation, BIS-guided anaesthesia and maintenance of optimal cerebral oxygen saturation will reduce cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* ASA 2-3 patients,
* > 18 years
* signed written consent for anesthesia and study participation
* Major abdominal surgery (stomach and intestin resection)
* epidural catheter insertion

Exclusion Criteria:

* pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Cognitive decline assessment change | three days
  Blood samples for determination of brain injury biomarkers (NSE, S 100, GFAP, TAU, UCH-L1, MMP-9, miRNA, apo E4) before and at the end of operation.
  Cognitive function testing (Mini mental test): before the operation and on day 2 after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alenka Spindler Vesel, MD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre, Ljubljana, Slovenia

REFERENCES:
- [Background] Pearse R, Dawson D, Fawcett J, Rhodes A, Grounds RM, Bennett ED. Early goal-directed therapy after major surgery reduces complications and duration of hospital stay. A randomised, controlled trial [ISRCTN38797445]. Crit Care. 2005;9(6):R687-93. doi: 10.1186/cc3887. Epub 2005 Nov 8. PMID 16356219
- [Background] Shoemaker WC, Appel PL, Kram HB, Waxman K, Lee TS. Prospective trial of supranormal values of survivors as therapeutic goals in high-risk surgical patients. Chest. 1988 Dec;94(6):1176-86. doi: 10.1378/chest.94.6.1176. PMID 3191758
- [Background] Green D, Paklet L. Latest developments in peri-operative monitoring of the high-risk major surgery patient. Int J Surg. 2010;8(2):90-9. doi: 10.1016/j.ijsu.2009.12.004. Epub 2010 Jan 14. PMID 20079469
- [Background] Wilson J, Woods I, Fawcett J, Whall R, Dibb W, Morris C, McManus E. Reducing the risk of major elective surgery: randomised controlled trial of preoperative optimisation of oxygen delivery. BMJ. 1999 Apr 24;318(7191):1099-103. doi: 10.1136/bmj.318.7191.1099. PMID 10213716
- [Background] Sandham JD, Hull RD, Brant RF, Knox L, Pineo GF, Doig CJ, Laporta DP, Viner S, Passerini L, Devitt H, Kirby A, Jacka M; Canadian Critical Care Clinical Trials Group. A randomized, controlled trial of the use of pulmonary-artery catheters in high-risk surgical patients. N Engl J Med. 2003 Jan 2;348(1):5-14. doi: 10.1056/NEJMoa021108. PMID 12510037
- [Background] Walsh SR, Tang T, Bass S, Gaunt ME. Doppler-guided intra-operative fluid management during major abdominal surgery: systematic review and meta-analysis. Int J Clin Pract. 2008 Mar;62(3):466-70. doi: 10.1111/j.1742-1241.2007.01516.x. Epub 2007 Nov 21. PMID 18031528
- [Background] Abbas SM, Hill AG. Systematic review of the literature for the use of oesophageal Doppler monitor for fluid replacement in major abdominal surgery. Anaesthesia. 2008 Jan;63(1):44-51. doi: 10.1111/j.1365-2044.2007.05233.x. PMID 18086070
- [Background] Gurgel ST, do Nascimento P Jr. Maintaining tissue perfusion in high-risk surgical patients: a systematic review of randomized clinical trials. Anesth Analg. 2011 Jun;112(6):1384-91. doi: 10.1213/ANE.0b013e3182055384. Epub 2010 Dec 14. PMID 21156979
- [Background] Giglio MT, Marucci M, Testini M, Brienza N. Goal-directed haemodynamic therapy and gastrointestinal complications in major surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Nov;103(5):637-46. doi: 10.1093/bja/aep279. PMID 19837807
- [Background] Slater JP, Guarino T, Stack J, Vinod K, Bustami RT, Brown JM 3rd, Rodriguez AL, Magovern CJ, Zaubler T, Freundlich K, Parr GV. Cerebral oxygen desaturation predicts cognitive decline and longer hospital stay after cardiac surgery. Ann Thorac Surg. 2009 Jan;87(1):36-44; discussion 44-5. doi: 10.1016/j.athoracsur.2008.08.070. PMID 19101265
- [Background] Chan MT, Cheng BC, Lee TM, Gin T; CODA Trial Group. BIS-guided anesthesia decreases postoperative delirium and cognitive decline. J Neurosurg Anesthesiol. 2013 Jan;25(1):33-42. doi: 10.1097/ANA.0b013e3182712fba. PMID 23027226
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Bisgaard J, Gilsaa T, Ronholm E, Toft P. Optimising stroke volume and oxygen delivery in abdominal aortic surgery: a randomised controlled trial. Acta Anaesthesiol Scand. 2013 Feb;57(2):178-88. doi: 10.1111/j.1399-6576.2012.02756.x. Epub 2012 Aug 17. PMID 22897633
- [Background] Brandstrup B, Tonnesen H, Beier-Holgersen R, Hjortso E, Ording H, Lindorff-Larsen K, Rasmussen MS, Lanng C, Wallin L, Iversen LH, Gramkow CS, Okholm M, Blemmer T, Svendsen PE, Rottensten HH, Thage B, Riis J, Jeppesen IS, Teilum D, Christensen AM, Graungaard B, Pott F; Danish Study Group on Perioperative Fluid Therapy. Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Ann Surg. 2003 Nov;238(5):641-8. doi: 10.1097/01.sla.0000094387.50865.23. PMID 14578723
- [Background] Holte K, Kehlet H. Fluid therapy and surgical outcomes in elective surgery: a need for reassessment in fast-track surgery. J Am Coll Surg. 2006 Jun;202(6):971-89. doi: 10.1016/j.jamcollsurg.2006.01.003. No abstract available. PMID 16735213
- [Background] Brandstrup B, Svendsen PE, Rasmussen M, Belhage B, Rodt SA, Hansen B, Moller DR, Lundbech LB, Andersen N, Berg V, Thomassen N, Andersen ST, Simonsen L. Which goal for fluid therapy during colorectal surgery is followed by the best outcome: near-maximal stroke volume or zero fluid balance? Br J Anaesth. 2012 Aug;109(2):191-9. doi: 10.1093/bja/aes163. Epub 2012 Jun 17. PMID 22710266
- [Background] Lobo SM, Ronchi LS, Oliveira NE, Brandao PG, Froes A, Cunrath GS, Nishiyama KG, Netinho JG, Lobo FR. Restrictive strategy of intraoperative fluid maintenance during optimization of oxygen delivery decreases major complications after high-risk surgery. Crit Care. 2011;15(5):R226. doi: 10.1186/cc10466. Epub 2011 Sep 23. PMID 21943111
- [Result] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Result] Sessler DI, Sigl JC, Kelley SD, Chamoun NG, Manberg PJ, Saager L, Kurz A, Greenwald S. Hospital stay and mortality are increased in patients having a "triple low" of low blood pressure, low bispectral index, and low minimum alveolar concentration of volatile anesthesia. Anesthesiology. 2012 Jun;116(6):1195-203. doi: 10.1097/ALN.0b013e31825683dc. PMID 22546967